CLINICAL TRIAL: NCT02535481
Title: A Multi-centre Randomised Controlled Trial to Compare Epidermal Grafting With Split Skin Grafting for Wound Healing
Brief Title: Epidermal Grafting in Wound Healing
Acronym: EPIGRAAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/0079
Record Dates: First submitted 2015-08-11; First posted 2015-08-28 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Ulcer; Skin Ulcer; Wounds and Injuries
Keywords: epidermal graft; suction blister; blister graft; suction graft; Epidermis/su, tr [Surgery, Transplantation]
MeSH Terms: conditions — Ulcer; Skin Ulcer; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidermal Graft (Experimental): The Cellutome Epidermal Graft Harvesting System will be used to harvest epidermal grafts as per existing normal clinical practice.
  Interventions: Device: Epidermal grafting
- Split Thickness Skin Graft (Experimental): Split thickness skin graft will be harvested using air dermatome as per normal clinical practise.
  Interventions: Procedure: Split thickness skin grafting

INTERVENTIONS:
Device: Epidermal grafting — The Cellutome Epidermal Graft Harvesting System will be used to harvest epidermal grafts.
  Other Names: CelluTome
  Arms: Epidermal Graft
Procedure: Split thickness skin grafting — Split thickness skin grafting will be performed as per normal clinical practice.
  Arms: Split Thickness Skin Graft

SUMMARY:
Split thickness skin grafting is the normal standard of care for wound closure. However, this is an invasive procedure and associated with pain also there can be additional donor site morbidity. Epidermal grafting is an emerging clinical alternative that is gaining clinical practise. Epidermal grafting (EG) is an alternative method of autologous skin grafting that 'harvests' a finer layer of skin than traditional Split thickness skin grafting (SSG). This potentially results in less pain and reduced donor site morbidity but only delivers several cell layers to the wound so may be less effective at healing a wound. It is not known if EG is an effective alternative to SSG.

Further the mechanism to achieve wound healing may be different. EG promotes wound healing by expressing growth factors that accelerates wound healing and encourages keratinocyte migration. Whereas SSG is a transplant of several skin layers that integrated to the existing wound bed as a formal skin covering.

The investigators wish to compare these two clinical practises; epidermal grafting and split thickness skin grafting in wound healing. Further to undertake a translational study to investigate the mechanism by which each technique achieves wound healing.

DETAILED DESCRIPTION:
This study evaluates the efficacy of EG, as an alternative to current wound management therapy, SSG. In a pilot study carried out in our centre (unpublished data), the investigators noted that this technique offers a method of autologous skin harvesting with minimal or no pain and a scar free donor site. Moreover, complete wound epithelialisation was achieved while maintaining patient independence. Therefore, this device has the potential to save healthcare resources, by eliminating the need for theatre space and a hospital bed, and result in better Patient Reported Outcomes Measures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18-90
3. Wound measuring more than 1cm x 1cm and lesser than 5cm x 5cm (1% TBSA)
4. Wound with clean, healthy granulating bed, with minimal adherent slough
5. Patient understands and is willing to participate and can comply with weekly visits and follow-up regime

Exclusion Criteria:

1. Wound with active infection
2. Wound at plantar of the foot
3. Patients unsuitable for Split Skin Grafting
4. Previous history of excessive bleeding associated with surgical biopsies or trauma
5. Allergies to tegaderm (and other dressings used in the study)
6. Known uncontrolled Diabetes Mellitus, as measured by an HbA1c > 10%.
7. Presence of one or more medical conditions, including renal, hepatic, hematologic, active auto-immune or immune diseases that, would make the subject an inappropriate candidate for this ulcer healing study
8. Patient not fit for surgery (ASA classification > 4)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toby Richards, MD FRCS, Principal Investigator — University College, London; Afshin Mosahebi, MBBS FRCS PhD MBA, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hampstead NHS Trust Hospital, London, United Kingdom

REFERENCES:
- [Derived] Kanapathy M, Bystrzonowski N, Hachach-Haram N, Twyman L, Becker DL, Richards T, Mosahebi A. Lower donor site morbidity and higher patient satisfaction with epidermal grafting in comparison to split thickness skin grafting: A randomized controlled trial (EPIGRAAFT Trial). J Plast Reconstr Aesthet Surg. 2020 Aug;73(8):1556-1564. doi: 10.1016/j.bjps.2020.03.006. Epub 2020 Mar 16. PMID 32532631
- [Derived] Kanapathy M, Hachach-Haram N, Bystrzonowski N, Harding K, Mosahebi A, Richards T. Epidermal grafting versus split-thickness skin grafting for wound healing (EPIGRAAFT): study protocol for a randomised controlled trial. Trials. 2016 May 17;17(1):245. doi: 10.1186/s13063-016-1352-y. PMID 27185033

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 61 patients were screened for eligibility; 44 of them fulfilled the inclusion criteria and were randomized to the two study groups (EG and SSG) between October 2015 and September 2017. Participants were recruited at the Royal Free London NHS Foundation Trust Hospital.
Groups:
- Epidermal Graft: Epidermal grafting: The Cellutome Epidermal Graft Harvesting System was used to harvest epidermal grafts.
- Split Thickness Skin Graft: Split thickness skin grafting: Split thickness skin grafting was performed as per normal clinical practice.
Period: Overall Study
Arm/Group | Epidermal Graft | Split Thickness Skin Graft
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidermal Graft | Split Thickness Skin Graft | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (19.9) | 59 (18) | 58.7 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 13 | 17 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Wound size (cm^2) [Mean (Standard Deviation); unit: cm^2] | 12.7 (9.9) | 16.5 (11) | 14.6 (10.7)
Duration of wound (week) [Mean (Standard Deviation); unit: week] | 48.9 (75.4) | 7.86 (16.1) | 28.4 (58.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Wounds With Complete Healing
Description: Number of wounds with complete healing at 6 weeks
Time Frame: 6 weeks and 3 months
Measure: Number; unit: number of wounds
Units Other Than Participants: Number of wounds
Arm/Group | Epidermal Graft | Split Thickness Skin Graft
Number analyzed (Participants) | 22 | 22
Number analyzed (Number of wounds) | 22 | 22
number of wounds
  6 weeks | 9 | 13
  3 months | 16 | 20
Statistical Analysis 1: Comparison: Epidermal Graft vs Split Thickness Skin Graft; Test type: Superiority; p = 0.366, Fisher Exact — At 6 weeks
Statistical Analysis 2: Comparison: Epidermal Graft vs Split Thickness Skin Graft; Test type: Superiority; p = 0.24, Fisher Exact — At 3 months

2. Primary Outcome: Mean Time for Donor Site Healing
Description: Complete donor site healing was defined as 100% re-epithelialisation and not requiring further dressings
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Epidermal Graft | Split Thickness Skin Graft
Number analyzed (Participants) | 22 | 22
days | 4.86 [4.41 to 5.32] | 21.32 [15.65 to 26.99]
Statistical Analysis 1: Comparison: Epidermal Graft vs Split Thickness Skin Graft; Test type: Superiority; p < 0.0001, Log Rank; Kaplan-Meier analysis of cumulative wound healing followed by a log rank test

3. Secondary Outcome: Time for Wound Healing
Description: Complete wound healing was defined as 100% re-epithelialisation and not requiring further dressings
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: week
Arm/Group | Epidermal Graft | Split Thickness Skin Graft
Number analyzed (Participants) | 22 | 22
week | 7.81 [6.44 to 9.19] | 6.59 [5.29 to 7.89]
Statistical Analysis 1: Comparison: Epidermal Graft vs Split Thickness Skin Graft; Test type: Superiority; p = 0.12, Log Rank

4. Secondary Outcome: Donor Site Morbidity
Description: The donor site morbidity was measured using the Vancouver Scar Scale (VSS). Total score scale ranges from 0 to 13. Lower score is more desirable as it represents a scar resembling normal surrounding skin. The scale assesses 4 categories: vascularity, height, pliability, and pigmentation. Total score is obtained by the sum of the categories.
Time Frame: 6 weeks and 3 months
Measure: Mean (Standard Deviation); unit: unit of a scale
Arm/Group | Epidermal Graft | Split Thickness Skin Graft
Number analyzed (Participants) | 22 | 22
unit of a scale
  6 weeks | 0.14 (0.45) | 3.73 (0.69)
  3 months | 0.09 (0.29) | 2.91 (0.67)
Statistical Analysis 1: Comparison: Epidermal Graft vs Split Thickness Skin Graft; Test type: Superiority; p = 0.001, t-test, 2 sided

5. Secondary Outcome: Patient Reported Outcome Measure (PROM)
Description: Patient reported outcome measure was assessed using a validated skin graft satisfaction questionnaire.The skin graft satisfaction questionnaire has a scale ranging from 1 to 7, with 1 representing very unsatisfied while 7 represents very satisfied. Hence, higher score represent higher satisfaction.
Time Frame: 6 weeks and 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Epidermal Graft | Split Thickness Skin Graft
Number analyzed (Participants) | 22 | 22
score on a scale
  6 weeks | 7 [7 to 7] | 6 [5 to 7]
  3 months | 7 [7 to 7] | 6 [6 to 7]
Statistical Analysis 1: Comparison: Epidermal Graft vs Split Thickness Skin Graft; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney) — At 6 weeks
Statistical Analysis 2: Comparison: Epidermal Graft vs Split Thickness Skin Graft; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney) — At 3 months

6. Secondary Outcome: Adverse Events
Description: Number of participants with of adverse events
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Epidermal Graft | Split Thickness Skin Graft
Number analyzed (Participants) | 22 | 22
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: The incidence of serious adverse events (SAEs) include mortality of any cause within the three months duration from the time of initial therapy, and the incidence of device-related adverse events (DAEs) and wound-related adverse events (WAEs) occurring within the study duration.
Arm/Group | Epidermal Graft | Split Thickness Skin Graft
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT02535481/Prot_SAP_000.pdf